CLINICAL TRIAL: NCT00001079
Title: Double-Blind Randomized Comparison Phase II Trial of Megestrol Acetate and Testosterone Enanthate in Combination Versus Megestrol Acetate Plus Testosterone Enanthate Placebo in Human Immunodeficiency Virus (HIV)-Associated Wasting.
Brief Title: A Study of Megestrol Acetate Alone or in Combination With Testosterone Enanthate Drug in the Treatment of HIV-Associated Weight Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 313; 11288 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; HIV Wasting Syndrome
Keywords: Placebos; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; HIV Wasting Syndrome; Megestrol Acetate; dihydrotestosterone heptanoate
MeSH Terms: conditions — HIV Infections; HIV Wasting Syndrome; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — testosterone enanthate; Megestrol Acetate

INTERVENTIONS:
Drug: Testosterone enanthate
Drug: Megestrol acetate

SUMMARY:
To test the hypothesis that the predominant accrual of fat rather than lean body mass (LBM) that occurs during treatment of HIV-associated wasting with megestrol acetate may be improved by treatment with megestrol acetate and testosterone enanthate in combination.

Body wasting is an increasingly frequent AIDS-defining condition in individuals infected with HIV. Increasing caloric intake fails to consistently restore lean tissue patients with HIV associated weight loss. Megestrol acetate has been shown to stimulate appetite and weight gain in subjects with cancer and in those with HIV associated weight loss. However, the weight gained during treatment with megestrol acetate was predominantly or exclusively fat. An important factor is the preferential increase in body fat seen in both of these studies may have been due to hypogonadism that occurs as a result of treatment with megestrol acetate, a progestational agent. Hypogonadism is associated with an increase in body fat and a decrease in LBM. Concomitant testosterone replacement should substantially increase the amount of LBM accrued during megestrol acetate therapy. This study will determine whether anabolic potential can be realized when caloric intake is increased in the absence of concomitant hypogonadism.

DETAILED DESCRIPTION:
Body wasting is an increasingly frequent AIDS-defining condition in individuals infected with HIV. Increasing caloric intake fails to consistently restore lean tissue patients with HIV associated weight loss. Megestrol acetate has been shown to stimulate appetite and weight gain in subjects with cancer and in those with HIV associated weight loss. However, the weight gained during treatment with megestrol acetate was predominantly or exclusively fat. An important factor is the preferential increase in body fat seen in both of these studies may have been due to hypogonadism that occurs as a result of treatment with megestrol acetate, a progestational agent. Hypogonadism is associated with an increase in body fat and a decrease in LBM. Concomitant testosterone replacement should substantially increase the amount of LBM accrued during megestrol acetate therapy. This study will determine whether anabolic potential can be realized when caloric intake is increased in the absence of concomitant hypogonadism.

This is a 24 week study consisting of a 12 week double blind, randomized comparison Phase II trial of megestrol acetate and testosterone enanthate in combination versus megestrol acetate plus testosterone enanthate placebo in HIV associated wasting and a 12 week open label follow up of the combination therapy.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Stable antiretroviral therapy provided the patient has been on it for >=30 days prior to study entry. AS PER AMENDMENT 9/26/97: Optimized antiretroviral therapy as determined by primary care provider with at least 30 days since initiation of such therapy.
* Standard maintenance and prophylaxis therapy for opportunistic infections is permitted provided patients have been on a stable dosage regimen for 2 weeks prior to screening.
* G-CSF.
* Erythropoietin.
* Any symptomatic therapy (e.g., analgesics, antihistamines, antiemetic, antidiarrheal agents, etc.).
* Replacement levels of thyroid drugs (same drug and dose as at 30 days pre-entry).
* Maintenance therapy is permitted for chronic opportunistic infections, but patient must be on a stable regimen for 14 days pre-entry.
* AS PER AMENDMENT 9/26/97: Oral nutritional supplements, dronabinol, cyproheptadine, or pentoxifylline.

Patients must have:

* Documented HIV-1 infection.
* Documented weight loss of > 10% pre-illness weight or Body Mass Index < 18.5 kg/m2. AS PER AMENDMENT 9/26/97: Documented weight loss of >= 5% pre-illness weight or Body Mass Index < 20 kg/m2.
* Life expectancy of at least 6 months.

NOTE:

* This protocol meets federal requirements governing prisoner participation in clinical trials.

Prior Medication:

Allowed:

* Stable (no change in drugs or dosage) antiretroviral therapy or no antiretroviral medications for >= 30 days prior to the study entry.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms or conditions are excluded:

* Diabetes mellitus.
* Diarrhea defined as 4 or more liquid or watery stools per day while using antidiarrheal medication.
* Tube feeding. AS PER AMENDMENT 9/26/97: Total or partial parenteral nutrition delivered centrally or peripherally.
* Impaired oral intake due to mucositis of any cause.
* Grade 2 or greater intractable nausea and vomiting despite medication.
* Cardiomyopathy or congestive heart failure.
* Persistent palpable dominant breast mass at study entry that has not been worked up - males and females.

Female patients:

* Pap smear or cervical biopsy that demonstrates high grade squamous intraepithelial lesions or cervical intraepithelial lesions 2 or worse.

Concurrent Medication:

Excluded:

* Systemic chemotherapy for B-cell lymphoma or malignancies other than Kaposi's sarcoma. (Patients with Kaposi's sarcoma receiving systemic chemotherapy will not be excluded.)
* Total or peripheral parenteral nutrition (oral supplements are not excluded).
* Anticoagulant therapy.
* Any drug that is designed to affect appetite or weight gain. AS PER AMENDMENT 9/26/97: Initiation of any new therapy designed to promote weight gain.
* Any change of antiretroviral or any change in the dosage of antiretroviral/s that had not been started 30 days pre-entry. AS PER AMENDMENT 9/26/97: Initiation of antiretroviral therapy within 12 weeks of protocol therapy for patients not previously receiving antiretroviral therapy.
* Anabolic hormones.
* Systemic glucocorticoids.
* Cytokine inhibitors.
* Oral contraceptives.
* Cytokines.
* Ketoconazole.
* Any other medication that might interfere with the objectives of this study.
* AS PER AMENDMENT 9/26/97:DHEA.

Patients with the following prior conditions will be excluded:

* Acute systemic opportunistic infections within 30 days prior to entry.
* Weight gain >= 3% as documented by self reporting or clinical records during the preceding 4 weeks. AS PER AMENDMENT 9/26/97: Enrollment of such patients should be deferred until weight stabilizes.
* History of hypersensitivity reaction to megestrol acetate or testosterone enanthate.
* History of cardiomyopathy or congestive heart failure.

Female patients:

* History of invasive cervical cancer.
* AS PER AMENDMENT 9/26/97: History of thromboemboli.

Prior Medication:

Excluded:

* No testosterone treatment within the previous 8 weeks.

Excluded within 30 days prior to entry:

* Ketoconazole.
* Initiation or change in antiretroviral therapy.
* Interleukins.
* Interferon, anabolic, hormonal or experimental therapies designed to improve appetite or weight gain (e.g., thalidomide, dronabinol, megestrol acetate, cyproheptadine, anabolic steroids, systemic glucocorticoids, pentoxifylline, or growth hormone).
* AS PER AMENDMENT 9/26/97: Dehydroepiandrosterone (DHEA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Schambelan M, Study Chair; Mulligan K, Study Chair; Von Roenn JH, Study Chair
Locations (21):
- United States (21):
  - USC CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Ucsf Aids Crs, San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Howard University Hosp., Div. of Infectious Diseases, ACTU, Washington D.C., District of Columbia
  - Queens Med. Ctr., Honolulu, Hawaii
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Indiana Univ. School of Medicine, Wishard Memorial, Indianapolis, Indiana
  - Tulane Med. Ctr. - Charity Hosp. of New Orleans, ACTU, New Orleans, Louisiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - Cornell University A2201, New York, New York
  - Memorial Sloan-Kettering Cancer Ctr., New York, New York
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Schambelan M, Zackin R, Mulligan K, Sattler FR, Chesney M, Stevens M, Edwards L, Egorin MJ, Von Roenn JH. Effect of testosterone (T) on the response to megesterol acetate (MA) in patients with HIV-associated wasting: a randomized, double-blind placebo-controlled trial (ACTG 313). 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 640)